CLINICAL TRIAL: NCT01805752
Title: Optimizing Integrated PMTCT Services in Rural North-Central Nigeria: A Cluster Randomized Trial
Brief Title: Optimizing Integrated PMTCT Services in Rural North-Central Nigeria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Muktar Aliyu, Assistant Professor of Preventive Medicine, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01HD075075-01 (NIH)
Record Dates: First submitted 2013-03-04; First posted 2013-03-06 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Suspected Damage to Fetus From Viral Disease in the Mother; HIV
Keywords: Prevention of mother to child HIV transmission; HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Integrated family-focused PMTCT arm (Experimental): Intervention package includes: 1) task-shifting to lower-cadre providers at PMTCT sites; 2) POC CD4+ cell count testing; (3) integrated mother-infant care; and (4) a prominent role for influential family members (male partners), working in close partnership with community-based health workers/volunteers.
  Patients attending sites randomized to this arm will also receive group health education; opt-out HIV testing, same-day HIV test results; infant feeding counseling; HBC services; infant prophylaxis, early infant diagnosis, and linkage to family spacing services, if desired.
  Interventions: Other: Task-shifting to lower-cadre providers at PMTCT sites; Other: POC CD4+ cell count testing; Other: integrated mother-infant care; Other: Prominent role for influential family members (male partners) in collaboration with CHWs
- Standard of care (No Intervention): Arm will receive standard of care activities, namely: group health education; opt-out HIV testing, same-day HIV test results; infant feeding counseling; HBC services; infant prophylaxis, early infant diagnosis, linkage to family spacing services, if desired.

INTERVENTIONS:
Other: Task-shifting to lower-cadre providers at PMTCT sites
  Arms: Integrated family-focused PMTCT arm
Other: POC CD4+ cell count testing
  Arms: Integrated family-focused PMTCT arm
Other: integrated mother-infant care
  Arms: Integrated family-focused PMTCT arm
Other: Prominent role for influential family members (male partners) in collaboration with CHWs
  Arms: Integrated family-focused PMTCT arm

SUMMARY:
Each year, an estimated 230,000 HIV-infected women in need of services for prevention of mother-to-child transmission of HIV (PMTCT) give birth in Nigeria, more than in any other nation in the world. Vanderbilt University (VU), through its affiliate, Friends in Global Health (FGH), is currently supporting HIV/AIDS services in North-Central Nigeria. These sites are predominantly rural primary health centers (PHCs) where shortages of high-cadre health care providers and insufficient laboratory capacity to perform CD4+ cell count testing have been major barriers to effective PMTCT scale-up. A systematic reassignment of patient care responsibilities coupled with the adoption of point-of-care (POC) CD4+ cell count testing will facilitate the ability of lower-cadre health providers to manage PMTCT care, including the provision and scale-up of antiretroviral treatment (ART) to pregnant women in these rural, decentralized sites. A system wherein men are facilitated to accompany their wives to ANC appointments will create an important opportunity to address entrenched gender norms. The investigators therefore propose using community and facility-based measures to encourage male partners to accompany their spouses for ANC. As influential community members, male partners can assist their spouses to utilize culturally-sensitive, sustainable and integrated PMTCT care provided by lower-cadre providers in these resource-constrained settings.

The investigators propose a parallel, cluster randomized trial to evaluate the impact of a family-focused PMTCT package that includes: 1) task-shifting to lower-cadre providers at PMTCT sites; 2) POC CD4+ cell count testing; (3) integrated mother-infant care; and (4)) a prominent role for influential family members (male partners), working in close partnership with community-based health workers/volunteers. The specific aims of this study are:

1. To evaluate whether implementation of the integrated PMTCT package in primary level antenatal clinics (ANC) increases the proportion of eligible pregnant women who initiate antiretroviral medications for the purposes of PMTCT. The investigators hypothesize that the provision of the PMTCT package in intervention clinics will improve PMTCT antiretroviral uptake rates among eligible women during pregnancy from 40% to 65%.
2. To determine whether implementation of the PMTCT package improves postpartum retention of mother-infant pairs at 6 and 12 weeks. The investigators hypothesize that postpartum retention rates among mother-infant pairs attending intervention sites will be >20% higher at 6 weeks when compared to mother-infant pairs receiving care in non-intervention sites.
3. Conduct a cost-effectiveness analysis (CEA) of the impact of this novel PMTCT intervention compared to the existing standard-of-care referral model. The investigators hypothesize that the proposed intervention will be more cost-effective than the existing model of care.

In addition, two qualitative evaluations will be conducted in order to:

1. Assess client satisfaction with health services, comparing PMTCT services provided by lower level vs. higher level cadre health workers; and
2. Evaluate health care worker satisfaction with the new PMTCT service delivery model.

DETAILED DESCRIPTION:
The investigators propose a parallel cluster randomized trial to evaluate the effects of the intervention. Twelve primary and secondary level health care facilities in Niger State will be randomized to the control (standard-of-care) or intervention arms. The investigators will match clinics on patient volume and level of facility and randomize to intervention and standard-of-care/control arms - 6 clinics per arm.

The investigators will make the proposed intervention available to all eligible women attending clinics that are randomized to the intervention arm. The drug regimens and general HIV care services provided as part of the package are standard of care, based on Nigerian national guidelines.

Inclusion Criteria: (1) HIV-infected women (and their infants) who present to ANC or delivery with unknown HIV status; (2) HIV-infected women (and their infants) with previous history of ARV prophylaxis or treatment, but who are not on prophylaxis or treatment at the time of presentation for antenatal care or delivery.

Exclusion Criteria: HIV-infected women with known status who are on ARV prophylaxis or treatment at the time of presentation to ANC.

Home-based care (HBC) workers will track clients who miss appointments at control and intervention sites. The HBC workers will document clients as terminated care if they: (1) discontinued services due to death or personal decision; (2) transferred their care to another clinic; or (3) are lost to follow-up (defined as being 90 days late for a clinic appointment plus 5 failed attempts at tracking the client). Clients will not receive any remuneration for participating in the study. Clients will be allowed to discontinue participation and decide that their medical data cannot be used in the analysis.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-infected women (and their infants) who present to ANC or delivery with unknown HIV status;
2. HIV-infected women (and their infants) with previous history of ARV prophylaxis or treatment, but who are not on prophylaxis or treatment at the time of presentation for antenatal care or delivery.

Exclusion Criteria:

HIV-infected women with known status who are on ARV prophylaxis or treatment at the time of presentation to ANC.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Proportion of eligible pregnant women who initiate ART for purposes of PMTCT | 18 months
  The primary outcome is the proportion of eligible women who initiate ARV medications for PMTCT. This will be determined through data in our electronic medical records system. The investigators will report the total proportion of women who initiate ARV drugs, presenting the results stratified by regimen (cART, ZDV, NVP) and type of facility. The investigators will also collect information on duration of cART.

SECONDARY OUTCOMES:
Postpartum retention of mother-infant pairs at 6 and 12 weeks post delivery | 12 weeks
  Mother-infant pairs who have presented for their 6-week postpartum appointment will be considered active in the program (retained in care). The investigators will assess retention at both 6 week and 12-week time points in order to examine the impact of our intervention package on early (6 week) and later (12-week) postpartum retention.

OTHER OUTCOMES:
HIV-free infant survival at 6 weeks postpartum | 6 weeks post delivery
  The study is not adequately powered to test this outcome.
Cost effectiveness analysis of impact of integrated PMTCT package | 18 months
  For the CEA, the basic outcome is the cost-effectiveness ratio (CER). The CER will be computed for both intervention and the standard-of-care arms.
  The investigators will also measure the incremental cost-effectiveness ratio (ICER). A separate ICER will be calculated for the two primary study outcomes (the cost/HIV-infected women who initiated treatment for PMTCT and the cost/mother-infant pair retained in care at 6 weeks postpartum) and for the secondary outcome (cost per infant infection averted at 6 weeks of age).

CONTACTS AND LOCATIONS:
Overall Officials: Muktar H Aliyu, MBBS, DrPH, Principal Investigator — Vanderbilt University
Locations (12):
- Nigeria (11):
  - CHC Agwara, Agwara, Niger State
  - Rural Hospital, Auna, Niger State
  - MCH Chanchaga, Chanchaga, Niger State
  - NCWS Farin Doki, Farin Doki, Niger State
  - BHC Garam, Garam, Niger State
  - PHC Gauraka, Gauraka, Niger State
  - BHC Ijah, Ijah, Niger State
  - BHC Izom, Izom, Niger State
  - Rural Hospital, Kaffin Koro, Niger State
  - MCH Paiko, Paiko, Niger State
  - BHC Wuse, Sabon Wuse, Niger State
- Rural Hospital, Aguié, Agaie, Niger

IPD SHARING:
Plan to Share IPD: No
IPD will not be available to other researchers.

REFERENCES:
- [Background] Aliyu MH, Blevins M, Audet C, Shepherd BE, Hassan A, Onwujekwe O, Gebi UI, Kalish M, Lindegren ML, Vermund SH, Wester CW. Optimizing PMTCT service delivery in rural North-Central Nigeria: protocol and design for a cluster randomized study. Contemp Clin Trials. 2013 Sep;36(1):187-97. doi: 10.1016/j.cct.2013.06.013. Epub 2013 Jun 29. PMID 23816493
- [Derived] Aliyu MH, Blevins M, Audet CM, Kalish M, Gebi UI, Onwujekwe O, Lindegren ML, Shepherd BE, Wester CW, Vermund SH. Integrated prevention of mother-to-child HIV transmission services, antiretroviral therapy initiation, and maternal and infant retention in care in rural north-central Nigeria: a cluster-randomised controlled trial. Lancet HIV. 2016 May;3(5):e202-11. doi: 10.1016/S2352-3018(16)00018-7. Epub 2016 Feb 24. PMID 27126487
- Available data/document: Clinical Study Report: doi: 10.1016/S2352-3018(16)000 — https://www.ncbi.nlm.nih.gov/pubmed/27126487 — Aliyu MH, Blevins M, Audet CM, Kalish M, Gebi UI, Onwujekwe O, Lindegren ML, Shepherd BE, Wester CW, Vermund SH. Integrated prevention of mother-to-child HIV transmission services, antiretroviral therapy initiation, and maternal and infant retention in care in rural north-central Nigeria: a cluster-randomised controlled trial. Lancet HIV. 2016 May;3(5):e202-11. doi: 10.1016/S2352-3018(16)00018-7. PubMed PMID: 27126487; PubMed Central PMCID: PMC4852280.